CLINICAL TRIAL: NCT01205438
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Subcutaneous LY2127399 in Patients With Systemic Lupus Erythematosus (SLE)
Brief Title: A Study of LY2127399 in Participants With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13653; H9B-MC-BCDT (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Results first posted 2018-06-19 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Systemic Lupus Erythematosus; Connective Tissue Disease; Autoimmune Disease
Keywords: SLE; Systemic Lupus Erythematosis; Lupus; autoimmune disease; LY2127399; Immune System Disease
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Connective Tissue Diseases; Autoimmune Diseases; Immune System Diseases | interventions — tabalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LY2127399 every 2 weeks (Experimental)
  Interventions: Drug: LY2127399
- LY2127399 every 4 weeks (Experimental): During the Treatment Period, for blinding purposes, participants will alternate injections of LY2127399 and injections of placebo every 2 weeks.
  Interventions: Drug: LY2127399; Drug: Placebo every 4 weeks
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo every 2 weeks

INTERVENTIONS:
Drug: LY2127399 — 120mg administered via subcutaneous injection for 52 weeks. 240 mg loading dose will be administered as the first dose of study drug
  Arms: LY2127399 every 2 weeks; LY2127399 every 4 weeks
Drug: Placebo every 2 weeks — Administered via subcutaneous injection for 52 weeks. A matching loading dose will also be administered at the first dose.
  Arms: Placebo
Drug: Placebo every 4 weeks — Administered via subcutaneous injection for 52 weeks.
  Arms: LY2127399 every 4 weeks

SUMMARY:
The purpose of this SLE study is to evaluate the efficacy, safety and tolerability of two different doses of LY2127399 administered in addition to standard of care therapy in participants with active SLE.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of SLE as defined by American College of Rheumatology (ACR) criteria
* Have positive antinuclear antibodies (ANA)
* Agree not to become pregnant throughout the course of the trial
* Have a screening SELENA-SLEDAI score ≥6. (The participant must be actively exhibiting all the symptoms scored on the screening SELENA-SLEDAI on the day of screening.)

Exclusion Criteria:

* Have active severe Lupus kidney disease
* Have active Central Nervous System or peripheral neurologic disease
* Have received intravenous immunoglobulin (IVIg) within 180 days of randomization
* Have active or recent infection within 30 days of screening
* Have had a serious infection within 90 days of randomization
* Have evidence or test positive for Hepatitis B
* Have Hepatitis C
* Are human immunodeficiency virus (HIV) positive
* Have evidence of active or latent tuberculosis (TB)
* Presence of significant laboratory abnormalities at screening
* Have had a malignancy in the past 5 years, except for cervical carcinoma in-situ or basal cell or squamous epithelial skin cell that were completely resected with no reoccurrence in the 3 yrs prior to randomization
* Have received greater than 40 mgs of prednisone or equivalent in the past 30 days
* Have changed your dose of antimalarial drug in the past 30 days
* Have changed your dose of immunosuppressive drug in the past 90 days
* Have previously received rituximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1124 (Actual)
Dates: Start 2011-01; Primary Completion 2014-08 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5PM Eastern time (UTC/GMT -5 hours, EST), Study Director — Eli Lilly and Company
Locations (183):
- United States (87):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anniston, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gilbert, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scottsdale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tempe, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malvern, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Covina, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., El Cajon, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Escondido, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Mesa, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lakewood, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Alamitos, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pasadena, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Riverside, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Gabriel, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Barbara, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Van Nuys, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Westlake Village, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Whittier, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aurora, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aventura, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., DeBary, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Naples, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Port Richey, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ormond Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pensacola, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pinellas Park, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plantation, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vero Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Duluth, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lithonia, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Meridian, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rockford, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Wayne, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Granger, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monroe, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Maine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cumberland, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Clair Shores, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Duluth, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hattiesburg, Mississippi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashua, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Freehold, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Voorhees Township, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Cruces, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albany, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brooklyn, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manhasset, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plainview, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roslyn, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chapel Hill, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Raleigh, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rocky Mount, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toledo, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Duncansville, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wyomissing, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cookeville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Knoxville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amarillo, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nassau Bay, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Round Rock, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Victoria, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St. George, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clarksburg, West Virginia
- Australia (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Leonards, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cairns, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maroochydore, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clayton, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malvern East
- Brazil (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Campinas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goiânia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Juiz de Fora
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto Alegre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salvador
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Canada (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamilton, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trois-Rivières, Quebec
- Ecuador (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cuenca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guayaquil
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Quito
- France (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orléans
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Strasbourg
- Hungary (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Debrecen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Győr
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gyula
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szeged
- India (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gujarat
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haryāna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabaad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kormangala
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pune
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trivandrum
- Israel (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haifa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kfar Saba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Petah Tikva
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Litwinsky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ẕerifin
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Riga, Latvia
- Malaysia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kota Kinabalu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kuala Lumpur
- Mexico (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mérida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Luis
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Luis Potosí City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tijuana
- New Zealand (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamilton
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Otahuhu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Takapuna
- Romania (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brasov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Galati
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Târgu Mureş
- Russia (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chelyabinsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kazan'
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kemerovo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orenburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tomsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yaroslavl
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yekaterinburg
- Serbia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belgrade
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kragujevac
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Niška Banja
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Novi Sad
- South Africa (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cape Town
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durban
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stellenbosch
- Spain (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., A Coruña
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bilbao
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Palmas de Gran Canaria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santiago de Compostela
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vigo
- Taiwan (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changhua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hualien City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaohsiung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
- Tunisia (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Marsa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monastir
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sfax
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sousse
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tunis
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tunis Monfleury
- United Kingdom (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cambridge, Cambridgeshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poole, Dorset
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Greater London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maidstone, Kent
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wigan, Lancashire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London

REFERENCES:
- [Derived] Vendel AC, Jaroszewski L, Linnik MD, Godzik A. B- and T-Lymphocyte Attenuator in Systemic Lupus Erythematosus Disease Pathogenesis. Clin Pharmacol Ther. 2024 Jul;116(1):247-256. doi: 10.1002/cpt.3282. Epub 2024 Apr 26. PMID 38676311
- [Derived] Toro-Dominguez D, Martorell-Marugan J, Martinez-Bueno M, Lopez-Dominguez R, Carnero-Montoro E, Barturen G, Goldman D, Petri M, Carmona-Saez P, Alarcon-Riquelme ME. Scoring personalized molecular portraits identify Systemic Lupus Erythematosus subtypes and predict individualized drug responses, symptomatology and disease progression. Brief Bioinform. 2022 Sep 20;23(5):bbac332. doi: 10.1093/bib/bbac332. PMID 35947992
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- [Derived] Li Y, Higgs RE, Hoffman RW, Dow ER, Liu X, Petri M, Wallace DJ, Dorner T, Eastwood BJ, Miller BB, Liu Y. A Bayesian gene network reveals insight into the JAK-STAT pathway in systemic lupus erythematosus. PLoS One. 2019 Dec 2;14(12):e0225651. doi: 10.1371/journal.pone.0225651. eCollection 2019. PMID 31790472
- [Derived] Kalunian KC, Urowitz MB, Isenberg D, Merrill JT, Petri M, Furie RA, Morgan-Cox MA, Taha R, Watts S, Silk M, Linnik MD. Clinical trial parameters that influence outcomes in lupus trials that use the systemic lupus erythematosus responder index. Rheumatology (Oxford). 2018 Jan 1;57(1):125-133. doi: 10.1093/rheumatology/kex368. PMID 29045736
- [Derived] Hoffman RW, Merrill JT, Alarcon-Riquelme MM, Petri M, Dow ER, Nantz E, Nisenbaum LK, Schroeder KM, Komocsar WJ, Perumal NB, Linnik MD, Airey DC, Liu Y, Rocha GV, Higgs RE. Gene Expression and Pharmacodynamic Changes in 1,760 Systemic Lupus Erythematosus Patients From Two Phase III Trials of BAFF Blockade With Tabalumab. Arthritis Rheumatol. 2017 Mar;69(3):643-654. doi: 10.1002/art.39950. PMID 27723281
- [Derived] Rovin BH, Dooley MA, Radhakrishnan J, Ginzler EM, Forrester TD, Anderson PW. The impact of tabalumab on the kidney in systemic lupus erythematosus: results from two phase 3 randomized, clinical trials. Lupus. 2016 Dec;25(14):1597-1601. doi: 10.1177/0961203316650734. Epub 2016 May 24. PMID 27220348
- [Derived] Merrill JT, van Vollenhoven RF, Buyon JP, Furie RA, Stohl W, Morgan-Cox M, Dickson C, Anderson PW, Lee C, Berclaz PY, Dorner T. Efficacy and safety of subcutaneous tabalumab, a monoclonal antibody to B-cell activating factor, in patients with systemic lupus erythematosus: results from ILLUMINATE-2, a 52-week, phase III, multicentre, randomised, double-blind, placebo-controlled study. Ann Rheum Dis. 2016 Feb;75(2):332-40. doi: 10.1136/annrheumdis-2015-207654. Epub 2015 Aug 20. PMID 26293163

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2127399 Every 2 Weeks: 120mg LY2127399 administered via subcutaneous injection for 52 weeks. 240 mg loading dose will be administered as the first dose of study drug.
- LY2127399 Every 4 Weeks: During the Treatment Period, for blinding purposes, participants will alternate injections of LY2127399 and injections of placebo every 2 weeks.
  120mg LY2127399 administered via subcutaneous injection for 52 weeks. 240 mg loading dose will be administered as the first dose of study drug
  Placebo every 4 weeks: Administered via subcutaneous injection for 52 weeks.
Period: Overall Study
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Weeks | Placebo
Started | 372 | 376 | 376
Received At Least One Dose of Study Drug | 371 | 374 | 376
Participated in Follow Up | 72 | 78 | 66
Completed | 295 | 289 | 288
Not Completed | 77 | 87 | 88
Not completed — Adverse Event | 19 | 17 | 24
Not completed — Death | 1 | 1 | 3
Not completed — Entry Criteria Not Met | 16 | 15 | 13
Not completed — Lack of Efficacy | 14 | 11 | 14
Not completed — Lost to Follow-up | 6 | 7 | 8
Not completed — Withdrawal by Subject | 19 | 25 | 19
Not completed — Physician Decision | 0 | 3 | 2
Not completed — Protocol Violation | 2 | 7 | 4
Not completed — Sponsor Decision | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Weeks | Placebo | Total
Number analyzed (Participants) | 372 | 376 | 376 | 1124
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (12.41) | 41.2 (12.73) | 41.9 (12.08) | 41.8 (12.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 342 | 346 | 349 | 1037
  Male | 30 | 30 | 27 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 110 | 92 | 99 | 301
  Not Hispanic or Latino | 229 | 233 | 235 | 697
  Unknown or Not Reported | 33 | 51 | 42 | 126
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 31 | 33 | 30 | 94
  Asian | 38 | 34 | 40 | 112
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 0 | 3
  Black or African American | 43 | 46 | 51 | 140
  White | 245 | 247 | 249 | 741
  More than one race | 14 | 14 | 6 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Ecuador | 20 | 17 | 12 | 49
  Russia | 12 | 19 | 12 | 43
  Romania | 9 | 8 | 13 | 30
  Hungary | 18 | 17 | 18 | 53
  United States | 143 | 137 | 148 | 428
  United Kingdom | 3 | 3 | 3 | 9
  Malaysia | 2 | 1 | 4 | 7
  India | 11 | 13 | 16 | 40
  Spain | 9 | 12 | 9 | 30
  New Zealand | 3 | 4 | 1 | 8
  Canada | 3 | 3 | 2 | 8
  Latvia | 3 | 4 | 2 | 9
  Taiwan | 20 | 14 | 16 | 50
  Brazil | 23 | 25 | 22 | 70
  Mexico | 19 | 22 | 23 | 64
  South Africa | 14 | 17 | 7 | 38
  Israel | 9 | 7 | 12 | 28
  Serbia | 19 | 25 | 32 | 76
  Australia | 9 | 7 | 3 | 19
  France | 2 | 1 | 1 | 4
  Tunisia | 21 | 20 | 20 | 61
Anti-dsDNA Antibody Level [Mean (Standard Deviation); unit: International Unit / Milliliter (IU/mL)] | 116.8 (118.17) | 110.6 (113.51) | 112.0 (116.60) | 113.1 (116.03)
Safety of Estrogens in Lupus Erythematosus National Assessment (SELENA-SLEDAI) Score [Mean (Standard Deviation); unit: units on a scale] — SELENA SLEDAI is calculated from 24 individual descriptors across 9 organ systems; 0 indicates inactive disease and the maximum theoretical score is 105; scores > 20 are rare.
  units on a scale | 10.4 (4.07) | 10.4 (4.17) | 9.8 (3.28) | 10.2 (3.86)
Physician's Global Assessment (PGA) Score [Mean (Standard Deviation); unit: units on a scale] — PGA is a single-item clinician rated assessment of the participant's current level of disease activity measured on a continuous 100-millimeter (mm) visual analytic scale with benchmarks of 0, 1, 2, and 3 from left to right corresponding to no, mild, moderate, and severe SLE disease activity.Scores are presented from 0 to 100. No worsening is defined as increase of ≥0.3 points.
  units on a scale | 47.2 (15.45) | 46.8 (15.60) | 44.9 (16.57) | 46.3 (15.90)
At Least One BILAG A or Two BILAG B Disease Activity Scores [Count of Participants; unit: Participants] — The British Isles Lupus Assessment Group (BILAG) instrument assesses global disease activity across 9 organ system domains. BILAG flare is assessed for each of the 9 organ domains using BILAG2004 index flare rules; A is a severe flare and B is a moderate flare.
  The sum of participants in all Categories for the Measure does not equal the Overall Number of Baseline Participants in the Arm/Group because not all participants will have at least one BILAG A or Two BILAG B Disease Activity scores.
  Participants | 230 | 218 | 209 | 657
Time of Onset of Lupus [Mean (Standard Deviation); unit: years] | 8.36 (8.500) | 7.94 (7.615) | 7.74 (7.078) | 8.01 (7.748)
Lupus Quality of Life (LupusQOL) Domain Scores [Mean (Standard Deviation); unit: units on a scale] — The LupusQoL is a disease-specific, 34-item, self-report questionnaire designed to measure the health-related quality of life (HRQoL) of participants with SLE within 8 domains.Responses are based on a 5-point Likert scale where 0 (all of the time) to 4 (never). A LupusQoL score for each domain is reported on a 0 to 100 scale, with greater values indicating better HRQoL. Population: All enrolled participants with LupusQOL baseline data.
  units on a scale
    Physical Health: number analyzed (Participants) | 366 | 364 | 365 | 1095
    Physical Health | 59.2 (24.98) | 59.1 (25.13) | 56.9 (26.17) | 58.4 (25.43)
    Emotional Health: number analyzed (Participants) | 366 | 364 | 365 | 1095
    Emotional Health | 65.7 (25.19) | 66.7 (23.99) | 64.6 (26.22) | 65.7 (25.14)
    Body Image: number analyzed (Participants) | 338 | 343 | 342 | 1023
    Body Image | 61.1 (28.99) | 63.2 (27.67) | 61.9 (29.20) | 62.1 (28.61)
    Pain: number analyzed (Participants) | 366 | 364 | 365 | 1095
    Pain | 56.1 (28.40) | 56.9 (26.75) | 53.6 (28.62) | 55.5 (27.95)
    Planning: number analyzed (Participants) | 366 | 364 | 365 | 1095
    Planning | 61.2 (30.37) | 62.1 (28.69) | 59.0 (30.92) | 60.8 (30.01)
    Fatigue: number analyzed (Participants) | 366 | 364 | 365 | 1095
    Fatigue | 56.0 (26.39) | 54.4 (25.54) | 53.4 (27.14) | 54.6 (26.36)
    Intimate Relationships: number analyzed (Participants) | 314 | 316 | 320 | 950
    Intimate Relationships | 56.2 (33.92) | 63.3 (31.53) | 56.8 (34.21) | 58.8 (33.36)
    Burden to Others: number analyzed (Participants) | 366 | 364 | 365 | 1095
    Burden to Others | 52.8 (30.70) | 51.9 (30.31) | 49.3 (32.39) | 51.3 (31.15)
Brief Fatigue Inventory (BFI) Score [Mean (Standard Deviation); unit: units on a scale] — BFI is a participants-reported scale that measures the severity of fatigue based on the worst fatigue experienced during the past 24-hours. The severity scores ranged from 0 (no fatigue) to 10 (fatigue as severe as you can imagine).
  units on a scale | 5.8 (2.57) | 5.6 (2.81) | 5.6 (2.81) | 5.6 (2.73)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving an SLE Responder Index Response at Week 52
Description: Percentage of participants with a ≥ 5 point reduction from baseline in SELENA SLEDAI score, and no worsening (increase of < 0.30 points from baseline) in PGA, and no new BILAG A organ domain score or 2 new BILAG B organ domain scores compared with baseline.
  SELENA SLEDAI is calculated from 24 individual descriptors across 9 organ systems; 0 indicates inactive disease and the maximum theoretical score is 105; scores > 20 are rare. PGA is a visual analog scale scored from 0 to 3 (0=none, 1=mild, 2=moderate, 3=severe). BILAG uses a single score for each of the 9 organ domains; range is from severe (A) to no disease (E). Participants who were unable to comply with allowed concomitant medications requirements were considered non-responders, as were participants who dropped out or were missing Week 52 data.
Time Frame: 52 weeks
Population: Intention to treat (ITT), all randomized participants who received at least one dose of study drug.Non-responder imputation (NRI) included.
Measure: Number; unit: percentage of participants
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Weeks | Placebo
Number analyzed (Participants) | 372 | 376 | 376
percentage of participants | 38.5 | 34.8 | 27.7

2. Secondary Outcome: Percentage of Participants Able to Decrease Dose of Prednisone or Equivalent With No Increase in Disease Activity at Week 52
Description: A participant achieves corticosteroid sparing effects (quiescent disease) if they have met the following criteria during Weeks 24 through 52; able to decrease their dose of prednisone or equivalent to 7.5 mg/day or less, have quiescent disease (BILAG C score or better in all nine systems), and no BILAG A or B flares in the previous three months, without an increase in either antimalarials or immunosuppressants on or prior to the visit.
Time Frame: 52 weeks
Population: Intention to treat (ITT), only participants receiving a prednisone or equivalent dose of more than 7.5 mg/day at baseline are included.
Measure: Number; unit: percentage of participants
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Weeks | Placebo
Number analyzed (Participants) | 146 | 129 | 131
percentage of participants | 21.2 | 14.7 | 11.5

3. Secondary Outcome: Change From Baseline to 52 Weeks in Anti-double Stranded Deoxyribonucleic Acid (Anti-dsDNA) Level
Description: Anti-double stranded deoxyribonucleic acid (anti-dsDNA) is a lab analyte used to assist in the diagnosis of SLE.
Time Frame: Baseline, 52 weeks
Population: Intention to treat (ITT), Last observation carried (LOCF). LOCF endpoint is defined as the latest post-baseline response obtained on or prior to the date of Week 52 or the date of early discontinuation from the treatment period.
Measure: Mean (Standard Deviation); unit: International Units (IU)
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Weeks | Placebo
Number analyzed (Participants) | 368 | 372 | 372
International Units (IU) | -27.7 (65.31) | -26.4 (64.13) | -7.0 (56.53)

4. Secondary Outcome: Change From Baseline to 52 Week Endpoint in Systemic Lupus Erythematosus Disease Activity Index (SLEDAI2K) Score
Description: SLE Disease Activity Index 2000 (SLEDAI-2K) score is a weighted, cumulative index of lupus disease activity. SLEDAI-2K is calculated from 24 individual descriptors across 9 organ systems; 0 indicates inactive disease and the maximum theoretical score is 105.
Time Frame: Baseline, 52 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Weeks | Placebo
Number analyzed (Participants) | 372 | 376 | 376
units on a scale
  Baseline | 10.3 (4.17) | 10.4 (4.01) | 9.8 (3.36)
  52 Weeks | -4.9 (4.57) | -4.7 (4.62) | -3.6 (4.21)

5. Secondary Outcome: Time to First Severe SLE Flare (SFI)
Description: The SFI uses the SELENA-SLEDAI disease activity index score, disease activity scenarios, treatment changes, and PGA to define mild/moderate and severe flares. The index takes into account the absolute change in total scores, new or worsening symptoms, and increases in corticosteroid use or hospitalization due to the disease activity.
  Time to first severe SLE flare (SFI) (in days) is calculated as: (Start date of first severe SLE flare (SFI) - Date of randomization + 1).
Time Frame: Baseline through 52 weeks
Population: Zero participants analyzed. Time to first severe SLE flare data was not collected for analysis.
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Weeks | Placebo
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Change From Baseline to 52 Week Endpoint in Physician's Global Assessment (PGA)
Description: PGA is a single-item clinician rated assessment of the participant's current level of disease activity measured on a continuous 100-millimeter (mm) visual analytic scale with benchmarks of 0, 1, 2, and 3 from left to right corresponding to no, mild, moderate, and severe SLE disease activity. Scores are presented from 0 to 100. No worsening defined as increase of ≤ 0.30 points from Baseline.
Time Frame: Baseline, 52 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Weeks | Placebo
Number analyzed (Participants) | 372 | 376 | 376
units on a scale | -21.2 (21.28) | -19.2 (23.13) | -15.1 (23.52)

7. Secondary Outcome: Change From Baseline to 52 Week Endpoint Lupus Quality of Life (LupusQOL) Domain Scores
Description: The LupusQoL is a disease-specific, 34-item, self-report questionnaire designed to measure the health-related quality of life (HRQoL) of participants with SLE within 8 domains.Responses are based on a 5-point Likert scale where 0 (all of the time) to 4 (never). A LupusQoL score for each domain is reported on a 0 to 100 scale, with greater values indicating better HRQoL.
Time Frame: Baseline, 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Weeks | Placebo
Number analyzed (Participants) | 372 | 376 | 376
units on a scale
  Physical Health: number analyzed (Participants) | 143 | 131 | 104
  Physical Health | 69.0 (26.42) | 66.2 (28.01) | 70.7 (27.78)
  Emotional Health: number analyzed (Participants) | 143 | 131 | 104
  Emotional Health | 72.7 (27.03) | 72.3 (27.72) | 74.0 (28.85)
  Body Image: number analyzed (Participants) | 139 | 128 | 97
  Body Image | 73.6 (27.79) | 72.8 (27.60) | 73.1 (29.76)
  Pain: number analyzed (Participants) | 143 | 131 | 104
  Pain | 68.5 (28.98) | 67.5 (29.78) | 71.4 (29.80)
  Planning: number analyzed (Participants) | 143 | 131 | 104
  Planning | 71.0 (30.04) | 70.7 (31.71) | 73.2 (33.39)
  Fatigue: number analyzed (Participants) | 143 | 131 | 104
  Fatigue | 65.5 (26.23) | 62.4 (28.17) | 69.3 (26.27)
  Intimate Relationships: number analyzed (Participants) | 132 | 118 | 95
  Intimate Relationships | 68.4 (33.39) | 66.1 (33.81) | 72.4 (31.42)
  Burden to Others: number analyzed (Participants) | 143 | 131 | 104
  Burden to Others | 62.6 (32.89) | 63.7 (31.06) | 69.2 (31.33)

8. Secondary Outcome: Percentage of Participants With No Worsening in Physician Global Assessment (PGA) Score at 52 Weeks
Description: Physician's Global Assessment (PGA) is a single-item clinician rated assessment of the participant's current level of disease activity measured on a continuous 100-mm visual analytic scale with benchmarks of 0, 1, 2, and 3 from left to right corresponding to no, mild, moderate, and severe SLE disease activity. Scores are presented from 0 to 100.No worsening defined as increase of ≤ 0.30 points from Baseline.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Weeks | Placebo
Number analyzed (Participants) | 372 | 376 | 376
percentage of participants | 32.8 | 37.8 | 42.8

9. Secondary Outcome: Change From Baseline to 52 Week Endpoint in Brief Fatigue Inventory (BFI) Scores
Description: A participants-reported scale that measures the severity of fatigue based on the worst fatigue experienced during the past 24-hours. The severity scores ranged from 0 (no fatigue) to 10 (fatigue as severe as you can imagine).
Time Frame: Baseline, 52 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Weeks | Placebo
Number analyzed (Participants) | 358 | 352 | 354
units on a scale | -0.7 (3.09) | -0.5 (2.91) | -0.5 (2.95)

10. Secondary Outcome: Time to First New British Isles Lupus Assessment Group (BILAG A) or 2 New BILAG B SLE Flares
Description: The British Isles Lupus Assessment Group (BILAG) instrument assesses global disease activity across 9 organ system domains. BILAG flare is assessed for each of the 9 organ domains using BILAG2004 index flare rules; A is a severe flare and B is a moderate flare.
  Time to first BILAG A or two BILAG B flares (in days) is calculated as: (Start date of first BILAG A or two BILAG B flares - Date of randomization + 1). The two BILAG B flares must occur in different domains at the same visit.
Time Frame: Baseline through 52 weeks
Population: Zero participants analyzed. Time to First New British Isles Lupus Assessment Group (BILAG A) or 2 New BILAG B SLE flare data was not collected for analysis.
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Weeks | Placebo
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Percentage of Participants With an Increase in Corticosteroids Dose at 52 Weeks
Description: An increase in corticosteroids at a visit was defined as a change from baseline greater than 2.5 mg/day in dose or prednisone or equivalent using average daily dose of corticosteroids taken since the previous scheduled visit.
Time Frame: 52 weeks
Population: Intention to treat (ITT), only participants receiving a prednisone or equivalent dose of more than 2.5 mg/day at baseline are included.
Measure: Number; unit: percentage of participants
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Weeks | Placebo
Number analyzed (Participants) | 295 | 289 | 288
percentage of participants | 4.7 | 6.2 | 5.9

12. Secondary Outcome: Change From Baseline to 52 Weeks Endpoint in SELENA-SLEDAI Disease Activity Score
Description: Safety of Estrogens in Lupus Erythematosus National Assessment - SLE Disease Activity Index (SELENA-SLEDAI) score is a weighted, cumulative index of lupus disease activity. SELENA-SLEDAI is calculated from 24 individual descriptors across 9 organ systems; 0 indicates inactive disease and the maximum theoretical score is 105.
Time Frame: Baseline, 52 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Weeks | Placebo
Number analyzed (Participants) | 368 | 367 | 372
units on a scale | -5.1 (4.62) | -4.8 (4.69) | -3.7 (4.31)

13. Secondary Outcome: Number of Participants With No New BILAG A and No More Than One New BILAG B Disease Activity Scores Compared to Baseline
Description: The British Isles Lupus Assessment Group (BILAG) instrument assesses global disease activity across 9 organ system domains. BILAG flare is assessed for each of the 9 organ domains using BILAG2004 index flare rules; A is a severe flare and B is a moderate flare.
Time Frame: Baseline through 52 weeks
Population: Intention to treat (ITT), all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Weeks | Placebo
Number analyzed (Participants) | 371 | 374 | 376
Participants | 134 | 144 | 160

14. Secondary Outcome: Percentage of Participants Achieving a Response as Measured by Modified SRI With No BILAG A or No More Than 1 BILAG B Organ Domain Flares at 52 Weeks
Description: Percentage of participants with a ≥ 5 point reduction from baseline in SELENA SLEDAI score, and no worsening (increase of < 0.30 points from baseline) in PGA, and no new BILAG A or no more than 1 new BILAG B organ domain flare compared with baseline. (Primary outcome modified to use BILAG flare instead of BILAG disease score)
  SELENA SLEDAI is calculated from 24 individual descriptors across 9 organ systems; 0 indicates inactive disease and the maximum theoretical score is 105. PGA is a visual analog scale scored from 0 to 3 (0=none, 1=mild, 2=moderate, 3=severe). BILAG flare is assessed for each of the 9 organ domains; A is a severe flare and B is a moderate flare. Participants who were unable to comply with allowed concomitant medications requirements were considered non-responders, as were participants who dropped out or were missing Week 52 data.
Time Frame: 52 weeks
Population: Intention to treat (ITT), all randomized participants who received at least one dose of study drug. Non-responder imputation (NRI) included.
Measure: Number; unit: percentage of participants
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Weeks | Placebo
Number analyzed (Participants) | 372 | 376 | 376
percentage of participants | 38.7 | 34.8 | 27.7

ADVERSE EVENTS:
Description: All participants who received at least 1 dose of study drug. For gender specific events, only occurring in male or female subjects, the number of subjects exposed has been adjusted accordingly.
Groups:
- LY2127399 Every 2 Weeks, Follow Up: 24-48 weeks post last dose for participants receiving LY2127399 every 2 weeks during the Treatment Period.
- LY2127399 Every 4 Wks, Follow Up: 24-48 weeks post last dose for participants receiving LY2127399 every 4 weeks during the Treatment Period.
- Placebo, Follow Up: 24-48 weeks post last dose for participants receiving placebo during the Treatment Period.
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Weeks | Placebo | LY2127399 Every 2 Weeks, Follow Up | LY2127399 Every 4 Wks, Follow Up | Placebo, Follow Up
Serious Adverse Events (participants affected / at risk) | 46/371 | 59/374 | 70/376 | 8/72 | 12/78 | 14/66
Other Adverse Events (participants affected / at risk) | 249/371 | 239/374 | 246/376 | 16/72 | 15/78 | 13/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2127399 Every 2 Weeks (N=371) | LY2127399 Every 4 Weeks (N=374) | Placebo (N=376) | LY2127399 Every 2 Weeks, Follow Up (N=72) | LY2127399 Every 4 Wks, Follow Up (N=78) | Placebo, Follow Up (N=66)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Addison's disease (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accommodation disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Serositis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lupus hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perinephric abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 2 (2) | 7 (7) | 1 (1) | 0 (0) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Salmonella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis syndrome (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic arthritis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Viral diarrhoea (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 6 (7) | 0 (0) | 0 (0) | 1 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of the vagina (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/341 (0) | 1/344 (1) | 0/349 (0) | 0/67 (0) | 1/74 (1) | 0/63 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/341 (0) | 0/344 (0) | 2/349 (2) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasculitis cerebral (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0/67 (0) | 0/74 (0) | 1/63 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Borderline personality disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysthymic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lupus nephritis (Renal and urinary disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obstructive uropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Renal mass (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urethral polyp (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0/341 (0) | 0/344 (0) | 1/349 (1) | 0 (0) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1/341 (1) | 0/344 (0) | 0/349 (0) | 0 (0) | 0 (0) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 0/341 (0) | 0/344 (0) | 1/349 (1) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0/341 (0) | 0/344 (0) | 1/349 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1/341 (1) | 0/344 (0) | 0/349 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 1/341 (1) | 0/344 (0) | 0/349 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lupus pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shrinking lung syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Butterfly rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Female sterilisation (Surgical and medical procedures) | 1/341 (1) | 0/344 (0) | 0/349 (0) | 0 (0) | 0 (0) | 0 (0)
Accelerated hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2127399 Every 2 Weeks (N=371) | LY2127399 Every 4 Weeks (N=374) | Placebo (N=376) | LY2127399 Every 2 Weeks, Follow Up (N=72) | LY2127399 Every 4 Wks, Follow Up (N=78) | Placebo, Follow Up (N=66)
Leukopenia (Blood and lymphatic system disorders) | 8 (8) | 4 (8) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 8 (8) | 9 (12) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 11 (16) | 13 (13) | 8 (9) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (6) | 9 (9) | 11 (13) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 25 (29) | 21 (30) | 32 (37) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 11 (14) | 5 (7) | 13 (16) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (8) | 7 (7) | 8 (8) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 23 (25) | 21 (24) | 35 (42) | 1 (1) | 3 (3) | 0 (0)
Toothache (Gastrointestinal disorders) | 9 (10) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 17 (21) | 9 (12) | 17 (20) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 8 (9) | 2 (3) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 11 (18) | 5 (7) | 12 (18) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 13 (16) | 6 (13) | 4 (8) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 9 (11) | 5 (14) | 5 (14) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 9 (35) | 13 (20) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Pyrexia (General disorders) | 7 (9) | 9 (11) | 8 (10) | 0 (0) | 0 (0) | 3 (3)
Bronchitis (Infections and infestations) | 18 (22) | 25 (29) | 22 (28) | 0 (0) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Conjunctivitis (Infections and infestations) | 4 (4) | 8 (8) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 7 (9) | 12 (14) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 10 (14) | 10 (10) | 13 (14) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 6 (7) | 10 (10) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 12 (15) | 17 (20) | 6 (7) | 0 (0) | 1 (2) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 9 (12) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 24 (28) | 18 (22) | 32 (41) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 4 (5) | 10 (14) | 5 (7) | 2 (2) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 11 (12) | 9 (9) | 18 (18) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 26 (26) | 27 (30) | 19 (23) | 2 (2) | 1 (1) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 5 (6) | 8 (8) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 58 (74) | 44 (60) | 45 (63) | 2 (2) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 53 (80) | 60 (81) | 63 (86) | 4 (6) | 3 (3) | 3 (4)
Vaginal infection (Infections and infestations) | 7/341 (9) | 5/344 (7) | 2/349 (2) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 9 (9) | 2 (2) | 6 (8) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 11 (13) | 5 (7) | 9 (18) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 2 (2) | 9 (10) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 8 (8) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (10) | 8 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (21) | 15 (16) | 15 (18) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 26 (27) | 21 (27) | 17 (20) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 4 (4) | 9 (9) | 2 (2) | 1 (1) | 2 (3) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 18 (19) | 12 (14) | 9 (9) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 9 (9) | 10 (10) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (8) | 10 (10) | 3 (5) | 0 (0) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 8 (8) | 11 (11) | 12 (12) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 34 (47) | 37 (50) | 34 (52) | 2 (2) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 8 (8) | 14 (17) | 8 (9) | 0 (0) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1/67 (1) | 0/74 (0) | 2/63 (2)
Anxiety (Psychiatric disorders) | 14 (15) | 11 (11) | 12 (12) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 14 (14) | 17 (18) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 13 (13) | 21 (22) | 15 (18) | 0 (0) | 3 (3) | 1 (1)
Penis disorder (Reproductive system and breast disorders) | 1/30 (1) | 0/30 (0) | 0/27 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 1/30 (1) | 0/30 (0) | 0/27 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (18) | 14 (14) | 17 (18) | 2 (2) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 10 (12) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 10 (11) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 8 (12) | 7 (7) | 8 (12) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 17 (17) | 8 (10) | 16 (16) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to product program termination, not all analyses were completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days